CLINICAL TRIAL: NCT06997861
Title: Parallel Randomized Study to Determine Pain Intensity and Quality of Life in Patients With Chronic Non-Cancer Pain Receiving Medication Review With Follow-up VS Usual Care
Brief Title: Medication Review Improves Pain Management and Quality of Life in Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polytechnic Institute of Porto (Other)
Collaborators: University of Salamanca (Other)
Responsible Party: Principal Investigator, Nuno Miguel da Silva Duarte, Principal Investigator, Polytechnic Institute of Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE/2023/87
Record Dates: First submitted 2025-05-18; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain
Keywords: Medication Review; Chronic Pain; Quality of Life; Pharmaceutical Care; Primary Care
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: single-blinded, randomized study
Who Masked: Participant
Masking Description: This trial is blinded to subjects. Each subject will be informed they will be allocated to one of the two arms without knowing which one. Subjects will know they will receive pharmaceutical care, despite not knowing what type of pharmaceutical care they will receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication Review (MR) (Experimental)
  Interventions: Other: Medication Review Type III
- Usual-Care (UC) (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Medication Review Type III — The MR arm will receive four MR interviews. In the first MR, information about the patient's personal and medical history, along with current health problems, relevant lab exams and medication will be gathered. This will be used to proceed with medication review process and assessment of Drug Related Problems (DRP) that may lead to negative medication results. A personalized care plan will be developed to correct any detected DRP, delivered in writing/e-mail to the patient and carefully explained. Some DRP's may need the physician's intervention to correct. In these cases, a detailed recommendation will be sent to the patient's physician via email. All physicians' recommendations acted upon or not, will be recorded. Subsequent interviews will assess patient compliance with the care plan and if necessary, adjustments will be made accordingly.
  Arms: Medication Review (MR)
Other: Usual Care — The UC arm will receive an intervention by the investigator at the same time frame defined for the MR arm. The intervention will also consist of interviews, although MR will not be conducted. The investigator will ask questions to the patient about is drug therapy in a similar fashion to what would happen in the community pharmacy. Simple advice and information will be carried out (i.e., reinforcement of adherence, explanation about indication of drugs etc.)
  Arms: Usual-Care (UC)

SUMMARY:
The goal of this parallel-group, single-blinded, randomized study is to conduct Medication Review (MR) Type III in chronic non-cancer pain patients to optimize drug therapy and measure it's influence on Pain Intensity and Quality of Life in the primary care setting. The study took place in Porto, Portugal with the collaboration of two Primary Care Units (USF Arca D'Água and USF Campanhã - Polo S. Roque da Lameira) under ACeS Porto Oriental, from where patients were recruited. The main question it aims to answer is:

* Does the implementation of pharmacist-led medication review benefit patients with chronic pain in the primary care setting?
* Researchers will compare with "Usual Care" (UC) patients which receives general advice on how to manage their pain and/or recommendations to take "over the counter" drugs, similar to community pharmacy visits, to see if there is a clinically significant difference in pain intensity and quality of life between the two groups of patients.
* Participants will be asked to attend face-to-face interviews once a month for 4 months with an expert in medication review, that evaluates their current medication and suggests an individualized care plan. These plans include measures aimed at physicians (e.g., medication adding; dose reduction) and participants (e.g., non-pharmacological measures; adherence to medication).

ELIGIBILITY:
Inclusion Criteria:

* Non-cancer chronic pain (>3 months, any cause)
* Follow-up at one of the selected Primary Care Units
* Average weekly pain score ≥4 at the screening phase
* Ability to attend monthly in-person or video interviews

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Dementia
* Other mental illness impairing self-reporting

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | From enrollment to the end of the interventions at 16 weeks
  Following IMMPACT recommendations, subjects will record weekly pain (defined as the average of three measurements in a week) scores in the following manner: In a 11-point NRS with three descriptors where 0 is "no pain", 5 is "moderate pain" and 10 "maximum pain", subjects will select which best describes the pain they felt in the last 24h and record their score in the morning. Also, subjects will be instructed to record their pain scores on the week previous to the interventions.

SECONDARY OUTCOMES:
Quality of Life (QoL) | From enrollment to the end of the interventions at 16 weeks
  In this study and according to the IMMPACT recommendations, the Brief Pain Inventory-short form (BPI) will be used to measure the pain interference using the interference scale of this QoL measurement instrument. Data regarding this outcome will be collected and registered in a similar fashion to PI. Patients will be instructed to fill out the BPI short form in paper in the same day they measure their third PI score.
Satisfaction with treatment | From enrollment to the end of the interventions at 16 weeks
  In accordance with IMMPACT recommendations, the Patient Global Impression of Change (PGIC) scale will be used to determine participants global satisfaction with interventions. The PGIC scale was adapted from the Clinical Global Impression scale, proposed for patients with schizophrenia. It is a unidimensional scale which consists of a 7-rating scale where 1 = "no change" up to 7 = "very much improved". Data regarding this outcome will be collected and registered in a similar fashion to primary outcomes. Patients will be instructed to fill out the PGIC on paper in the same day they measure their third PI score and BPI.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Investigação em Saúde e Ambiente (CISA) - School of Health of the Polytechnic Institute of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the study (including de-identified individual-level data) will be made available upon reasonable request. The data will include all variables used in the analysis relevant to the primary and secondary outcomes, excluding any information that could compromise participant privacy or confidentiality.
Supporting Information: Study Protocol, ICF
Time Frame: The IPD will be available beginning 6 months after publication of the primary results and will remain available for up to 4 years following publication.
Access Criteria: Researchers who provide a methodologically sound proposal and have appropriate institutional approval may request access. Proposals should be submitted to the study principal investigator via email. A data use agreement will be required prior to the release of data.

REFERENCES:
- [Background] McDermott ME, Smith BH, Elliott AM, Bond CM, Hannaford PC, Chambers WA. The use of medication for chronic pain in primary care, and the potential for intervention by a practice-based pharmacist. Fam Pract. 2006 Feb;23(1):46-52. doi: 10.1093/fampra/cmi068. Epub 2005 Aug 17. PMID 16107494
- [Background] Kadam P, Bhalerao S. Sample size calculation. Int J Ayurveda Res. 2010 Jan;1(1):55-7. doi: 10.4103/0974-7788.59946. No abstract available. PMID 20532100
- [Background] Domingues L, Cruz E. Adaptação Cultural e Contributo para a Validação da Escala Patient Global Impression of Change. Ifisionline. 2011;2(1):31-7
- [Background] Cleeland CS. The Brief Pain Inventory User Guide. University of Texas ; 2009
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen M. Further Validation of a Portuguese Version of the Brief Pain Inventory Interference Scale. Clin Salud. 2012;23(1):89-96
- [Background] Sabater Hernández D, Milena Castro Silva M, María Faus Dáder J. Método Dáder: manual de seguimento farmacoterapêutico. 3a. Lisboa: Edições Universitárias Lusófonas; 2009
- [Background] Wan X, Wang W, Liu J, Tong T. Estimating the sample mean and standard deviation from the sample size, median, range and/or interquartile range. BMC Med Res Methodol. 2014 Dec 19;14:135. doi: 10.1186/1471-2288-14-135. PMID 25524443
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] International Pharmaceutical Federation (FIP). International Pharmaceutical Federation (FIP). Medication review and medicines use review: A toolkit for pharmacists. The Hague: International Pharmaceutical Federation; 2022.
- [Background] Griese-Mammen N, Hersberger KE, Messerli M, Leikola S, Horvat N, van Mil JWF, Kos M. PCNE definition of medication review: reaching agreement. Int J Clin Pharm. 2018 Oct;40(5):1199-1208. doi: 10.1007/s11096-018-0696-7. Epub 2018 Aug 2. PMID 30073611
- [Background] Hepler CD, Strand LM. Opportunities and responsibilities in pharmaceutical care. Am J Hosp Pharm. 1990 Mar;47(3):533-43. PMID 2316538
- [Derived] Duarte N, Martins JP, Garcia-Domingo M, Garcia-Pedraza JA, Santos M. Medication review improves pain management and quality of life in chronic pain: a pilot randomized controlled study. Sci Rep. 2025 Dec 29;15(1):44689. doi: 10.1038/s41598-025-28475-8. PMID 41461687